CLINICAL TRIAL: NCT04891679
Title: A Randomised Control Study of Titrated and Static Oral Misoprostol for Induction of Labor at Term
Brief Title: Induction of Labor by Oral Misoprostol Solution
Acronym: OMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Responsible Party: Principal Investigator, Dr. Barbie Sharma, Senior Resident, Department of obstetrics and gynecology, Christian Medical College and Hospital, Ludhiana, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Titrated and Static OMS
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Induction of Labor

STUDY DESIGN:
Intervention Model Description: Single center interventional single-blinded randomised controlled trial
Who Masked: Participant
Masking Description: Women were randomized (1:1) into the treatment groups A) Titrated-dose OMS group B) Static dose OMS group; using computer generated number sequence. Allocation concealment was carried out by using opaque envelopes that were distributed by the obstetrics nurse. Whereas study investigators and attending care teams were aware of the allocated arm, patients were kept blinded to the allocation. Study investigators and outcome assessors could not be blinded as the data collection and analysis included outcome measures like timing of oral misoprostol solution doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Titrated OMS) (Active Comparator): Titrated oral misoprostol solution
  Interventions: Drug: Oral misoprostol solution (OMS)
- Group B (Static OMS) (Active Comparator): Static oral misoprostol solution
  Interventions: Drug: Oral misoprostol solution (OMS)

INTERVENTIONS:
Drug: Oral misoprostol solution (OMS) — Based on the WHO labor induction recommendation, and for the purpose of achieving precise oral misoprostol dosage, one misoprostol tablet (200 mcg) was pulverized and dissolved into 200 ml water.90 Thus 1ml of solution had 1mcg of misoprostol. This misoprostol solution could be preserved at room temperature and remained active for 24 hours.
  Hourly titrated oral misoprostol solution was given to group A as described by Wang X et al, 2016 as described below.
  0 hour= 20ml
  1. hour= 20ml
  2. hour= 30ml
  3. hour= 30ml
  4. hour= 30ml
  5. hour= 40ml 6.5 hour= 50ml 8.5 hour= 60ml 10.5 hour=60ml
  Group B received 25 mcg (25 ml) oral misoprostol solution every 2 hours for a maximum of 12 doses or until the onset of regular uterine activity.

SUMMARY:
AIM: To evaluate effectiveness and safety of titrated oral misoprostol solution (OMS) in comparison with static-dose oral misoprostol solution for induction of labor at term.

Women with singleton live pregnancy at term without any complications who were admitted in labor room for induction of labor were enrolled.

Study involves allocation of selected women in two groups randomly and use of either titrated or static oral misoprostol dose regimen to induce labor. Possible benefits included rapid induction of labor with oral drug regimen which is easier to comply as compared to vaginal regimens. Women were at risk of all the complications associated with induction of labor like labor abnormalities, risk of cesarean section, non reassuring fetal status.

DETAILED DESCRIPTION:
This comparative randomized study was conducted in the Department of Obstetrics and Gynecology, Christian medical college and hospital, Ludhiana for a period of one year beginning from 1st December, 2017 to 30th November, 2018. The study group comprised of all antenatal women admitted in labor room at term for induction of labor. Informed consent was taken for all selected women. Women were subjected to detailed history taking, a complete physical examination including per vaginum examination (to calculate modified bishop's score and to rule out cephalopelvic disproportion), investigations and a NST. Gestational age was established by the first date of the last menstrual period and confirmed by first trimester ultrasound. Presentation was confirmed by palpation and third trimester ultrasound.

Women after randomization were allocated into two groups. The first group (A) was induced with hourly titrated oral misoprostol regimen and the second group (B) received two hourly static oral misoprostol regimen. Once labor had started, vital signs were closely monitored every 2 hours; fetal heart rate (FHR) and uterine activity every 15 minutes during first stage of labor. Per vaginum examination was done 4-hourly or as indicated.

Primary and secondary outcome measures were noted and analyzed to compare safety and efficacy of titrated and oral misoprstol solution.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton live pregnancy;
2. ≥37 weeks gestation;
3. Cephalic presentation;
4. Reassuring fetal heart rate;
5. Modified Bishop'score

Exclusion Criteria:

1. Hypersensitivity to misoprostol;
2. Uterine scar due to previous cesarean section or other uterine surgery;
3. Grand multipara;
4. Multiple gestations;
5. High risk pregnanacies • preeeclampsia with severe features • significant maternal cardiac,renal, liver disease
6. Any contraindication to induction and vaginal delivery e.g. cephalopelvic disproportion, malpresentation, fetal compromise and ante partum hemorrhage
7. Intrauterine fetal demise

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant females were enrolled for induction of labor in the study.
Enrollment: 264 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Interval between induction and delivery | From first dose of oral misoprostol solution (titrated/static) to childbirth; upto 5 days
  The time taken from induction of labor to delivery measured as
  1) <12 hours 2) 12-24 hours 3) 24-48 hours 4) >48 hours

SECONDARY OUTCOMES:
Mean change in modified Bishop's score | From first dose of oral misoprostol solution to childbirth (intrapartum); upto 5 days
  Measured as difference between modified bishop's score before induction of labor and at amniotomy/stopping of oral misoprostol solution regimen; minimum 0f 1 to maximum of 7.
Number of misoprostol doses | From first dose of oral misoprostol solution to childbirth (intrapartum); upto 5 days
  Measured as 1-2; 3-4; 5-6; 7-8; >9
Time taken to give required doses | From first dose of oral misoprostol solution to childbirth (intrapartum); upto 5 days
  Measured as 1-4 hours; 5-8 hours; 9-12 hours; 13-16 hours; 17-20 hours; 21-24 hours
Total misoprostol dosage | From first dose of oral misoprostol solution to childbirth (intrapartum); upto 5 days
  Measured as </=75mcg; 76-150mcg; 151-225mcg; 226-300mcg; >301 mcg
Mode of delivery | Upto 5 days from first dose of oral misoprostol solution
  In terms of Vaginal delivery/LSCS
Indication for LSCS | Upto 5 days from first dose of oral misoprostol solution
  Divided into either of the following:
  1. SECONDARY ARREST OF DILATATION
  2. MSAF IN EARLY LABOR
  3. CTG CATEGORY III
  4. FAILED INDUCTION
  5. CEPHALOPELVIC DISPROPORTION
  6. CORD PROLAPSE
  7. DEEP TRANSVERSE ARREST
  8. ARREST OF DESCENT OF HEAD
Oxytocin augmentation | From first dose of oral misoprostol solution to childbirth (intrapartum); upto 5 days
  Required/Not required
Maternal morbidity | From first dose of oral misoprostol solution to dischage from hospital; upto 7 days
  In terms of incidence of either of the following:
  1. Incidence of tachysystole
  2. Fever- intrapartum and postpartum
  3. Puerperal sepsis
  4. Uterine rupture
Neonatal parameters | From childbirth to discharge of the baby; upto 1 month
  Measured in terms of incidence of either of the following:
  1. Incidence of meconium-stained liquor
  2. APGAR scores at 1,5 min
  3. NICU stay

CONTACTS AND LOCATIONS:
Overall Officials: SUNITA GOYAL, MBBS, MD, Study Chair — Department of obstetrics and gynecology, Christian Medical College and hospital, Ludhiana
Locations (1):
- Christian Medical College and Hospital, Ludhiana, Punjab, India

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in the study, after deidentification (text, tables, figures and appendices) will be shared in the excel sheet format.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning immediately and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data for any purpose. Link will be made available at a later date.

REFERENCES:
- [Background] Rouzi AA, Alsahly N, Alamoudi R, Almansouri N, Alsinani N, Alkafy S, Rozzah R, Abduljabbar H. Randomized clinical trial between hourly titrated and 2 hourly static oral misoprostol solution for induction of labor. Am J Obstet Gynecol. 2017 Apr;216(4):405.e1-405.e6. doi: 10.1016/j.ajog.2016.11.1054. Epub 2016 Dec 14. PMID 27986461
- [Background] Aduloju OP, Ipinnimo OM, Aduloju T. Oral misoprostol for induction of labor at term: a randomized controlled trial of hourly titrated and 2 hourly static oral misoprostol solution. J Matern Fetal Neonatal Med. 2021 Feb;34(4):493-499. doi: 10.1080/14767058.2019.1610378. Epub 2019 Apr 29. PMID 31006282
- Available data/document: Informed Consent Form: PATIENT INFORMATION SHEET — https://figshare.com/s/a6c10a2a4be65f30144b
- Available data/document: Study Protocol: STUDY PROTOCOL — https://figshare.com/s/3f978a10eee4e90173bb